CLINICAL TRIAL: NCT01219088
Title: Post Operative Pain Control Among Intrathecal 0.1 mg Morphine, Femoral Nerve Block, or Periarticular Infiltration of 20 mL of 0.25% Bupivacaine in Patients Post Intramedullary Hip Screw
Brief Title: Intrathecal Morphine,Femoral Nerve Block,Periarticular Bupivacaine Infiltration for Pain After Intramedullary Hip Screw
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Assoc. Prof. Thitima Chinachoti, M.D., Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si392/2010
Record Dates: First submitted 2010-09-15; First posted 2010-10-13 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Controlled group (No Intervention): Spinal anesthesia with 0.5% bupivacaine alone
  Interventions: Drug: Bupivacaine, morphine
- Femoral nerve block (Active Comparator): Spinal anesthesia plus femoral nerve block with 20 mL of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine, morphine
- Intrathecal morphine (Active Comparator): Spinal anesthesia plus 0.1 mg of intrathecal morphine
  Interventions: Drug: Bupivacaine, morphine
- Periarticular bupivacaine infiltration (Active Comparator): Spinal anesthesia plus periarticular infiltration with 20 mL of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine, morphine

INTERVENTIONS:
Drug: Bupivacaine, morphine — 1.8-2.5 mL of 0.5% heavy bupivacaine for spinal anesthesia 20 mL of 0.25% bupivacaine for femoral nerve block 0.1 mg of intrathecal morphine 20 mL of 0.25% bupivacaine for periarticular infiltration

SUMMARY:
Falls are a common problem in elderly patients resulting fractured femur, which require early operation. Adequate postoperative pain control will provide good recovery. The investigators will compare the efficacy of postoperative pain control among intrathecal morphine, femoral nerve block, and periarticular infiltration with bupivacaine in patients undergone intramedullary hip screw under spinal anesthesia.

DETAILED DESCRIPTION:
Study methods :

Every patients without any exclusion criteria will be performed spinal anesthesia by 0.5% heavy bupivacaine then divided into 4 groups

1. Controlled group : spinal anesthesia alone
2. Femoral nerve block by 20 mL of 0.25% bupivacaine before spinal anesthesia
3. Spinal anesthesia plus 0.1 mg morphine intrathecally
4. Spinal anesthesia plus periarticular infiltration with 20 mL of 0.25% bupivacaine

All patients will receive postoperative intravenous patient controlled analgesia (IV PCA) morphine for 48 hours.

Data collection

1. Demographic data
2. Pain score : preoperative, 3 hours postoperative in the 1st six hours, 12 hours postoperative by visual analog scoring system (VASS)
3. Patient global assessment and patient satisfactory VASS at 24 and 48 hours postoperative
4. The amount of morphine at 24 and 48 hours postoperative and the time of the 1st dose

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* good consciousness, well co-operated, can use PCA machine
* ASA class 1-3
* no contraindication of spinal anesthesia
* accept for spinal anesthesia
* body weight > 30 kg
* BMI 20-35 kg/m2
* no history of research-drug allergy

Exclusion Criteria:

* previous history of hip surgery (the same side)
* pathological fractured such as severe infection, bone cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The amount of morphine consumption. | 24 hours postoperative

SECONDARY OUTCOMES:
Efficacy of pain control | 48 hours postoperative
  Efficacy of pain control measured by
  1. The amout of morphine consumption
  2. Visual analogue pain scale
  3. Patient satisfaction by patient global assessment
  4. Incidences of adverse events : nausea, vomiting, pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Thitima Chinachoti, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043